CLINICAL TRIAL: NCT07354503
Title: The Efficacy and Safety of Telitacicept in the Treatment of Pediatric IgA Vasculitis-Associated Nephritis: A Multicenter Clinical Study
Brief Title: Telitacicept in the Treatment of Pediatric IgA Vasculitis-Associated Nephritis
Status: Not yet recruiting | Type: Observational
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Mao Jianhua, Director, Head of Nephrology, Principal Investigator, Clinical Professor, The Children's Hospital of Zhejiang University School of Medicine
Other Study IDs: TTPIgAVN
Record Dates: First submitted 2025-12-30; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: IgAVN; IgA Vasculitis
Keywords: IgAV nephritis; Telitacicept; Children
MeSH Terms: conditions — IgA Vasculitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 48 Weeks
Biospecimen Retention: Samples Without DNA — During the research process, it is necessary to collect peripheral blood and urine samples from the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

GROUPS / COHORTS (3):
- Glucocorticoids group: Throughout the treatment period, the participants were administered glucocorticoids but did not receive any immunosuppressants or biologic therapies.
  Interventions: Device: Collect clinical data from the patients.; Drug: This study exclusively prospectively collected clinical data from the patients and did not involve any therapeutic interventions
- Telitacicept group: Throughout the treatment period, the participants were administered telitacicept but did not receive any immunosuppressants, glucocorticoids and other biologic therapies.
  Interventions: Device: Collect clinical data from the patients.; Drug: This study exclusively prospectively collected clinical data from the patients and did not involve any therapeutic interventions
- Glucocorticoids combined Telitacicept group: Throughout the treatment period, the participants were administered both glucocorticoids and telitacicept but did not receive any immunosuppressants or other biologic therapies.
  Interventions: Device: Collect clinical data from the patients.; Drug: This study exclusively prospectively collected clinical data from the patients and did not involve any therapeutic interventions

INTERVENTIONS:
Device: Collect clinical data from the patients. — This study exclusively prospectively collected clinical data from the patients and did not involve any therapeutic interventions.
Drug: This study exclusively prospectively collected clinical data from the patients and did not involve any therapeutic interventions — This study exclusively prospectively collected clinical data from the patients and did not involve any therapeutic interventions

SUMMARY:
To further evaluate the efficacy and safety of Telitacicept in the treatment of pediatric IgA vasculitis nephritis (IgAVN) within real-world settings, this study employs a multicenter, retrospective and prospective observational research design. It aims to compare the efficacy of Telitacicept with that of glucocorticoids, thereby providing clinicians with a reference for the rational and standardized application of Telitacicept.

DETAILED DESCRIPTION:
IgA vasculitis (IgAV) is a common form of vasculitis in children, with an annual incidence ranging from 6.1 to 55.9 cases per 100,000 children. The highest incidence is observed in those aged 4 to 6 years. When the kidneys are affected, the condition is referred to as IgAV nephritis (IgAVN), impacting approximately 20% to 80% of children with IgAV, thus making it one of the most prevalent secondary glomerular diseases in this population. Most cases of childhood IgAVN are mild or self-limiting; however, a subset of children may experience severe renal involvement, which may manifest as nephrotic syndrome, significant proteinuria, elevated serum creatinine levels, hypertension, persistent proteinuria, and renal biopsy results indicating over 50% crescent involvement. Research indicates that among children with moderate to severe proteinuria due to IgAVN, approximately 10% to 20% may progress to end-stage renal disease (ESRD), with persistent proteinuria identified as an independent risk factor for poor prognosis in IgAVN. Currently, clinical management primarily relies on corticosteroids, calcineurin inhibitors (CNI), mycophenolate mofetil (MMF), cyclophosphamide (CTX), and other immunosuppressants. However, some children exhibit poor responses to conventional treatments, and prolonged use of these medications may lead to various adverse effects, including infections, metabolic disorders, and growth impairment.

The increased presence of galactose-deficient IgA1 (Gd-IgA1) in circulation is a critical factor in the pathogenesis of IgAVN. Gd-IgA1 serves as an antigen that binds to autoantibodies, resulting in the deposition of immune complexes in the mesangium of the glomeruli, mesangial proliferation, inflammation, and subsequent glomerular damage. Telitacicept is a transmembrane activator and calcium modulator and cyclophilin ligand interactor (TACI) fused protein that specifically binds to both B lymphocyte stimulator (BLys) and a proliferation-inducing ligand (APRIL), thereby inhibiting the maturation and differentiation of B lymphocytes, plasma cell formation, and antibody production. A multicenter retrospective clinical study of Telitacicept in children with refractory IgA nephropathy (IgAN) and IgAVN demonstrated a gradual decrease in proteinuria in both groups throughout the treatment period, with consistent trends observed. In the IgAVN subgroup, following treatment with Telitacicept for 4, 12, 24, 36, and 48 weeks, 24-hour urinary protein levels decreased by 65.1%, 77.2%, 91.2%, 84.7%, and 85.8%, respectively, compared to baseline, while the urine protein-to-creatinine ratio (UPCR) decreased by 41.3%, 65.4%, 77.9%, 82.2%, and 87.8%. Additionally, a study involving seven children with IgAVN reported a 68.3% reduction in average 24-hour urinary protein after 24 weeks of Telitacicept treatment, with stable estimated glomerular filtration rates (eGFR) maintained throughout the treatment period. Furthermore, another study indicated that after 24 weeks of Telitacicept treatment, urinary protein levels significantly decreased, and hematuria improved markedly. None of the three studies reported serious adverse events.

Despite these promising findings, the clinical application of Telitacicept in children with IgAVN is still in the early exploratory stage, based on small sample studies with limited clinical follow-up. To further assess the efficacy and safety of Telitacicept in treating pediatric IgAVN in real-world settings, this study employs a multicenter retrospective plus prospective observational research design to compare the efficacy of Telitacicept withglucocorticoids, aiming to provide a reference for clinicians regarding the rational and standardized application of Telitacicept.

ELIGIBILITY:
Inclusion Criteria:

1. Age 3-17 years;
2. Patients diagnosed with IgA vasculitis nephritis (IgAVN) based on clinical manifestations and renal pathological diagnosis;
3. Urinary protein quantification requirements: urinary protein/creatinine ratio (UPCR) of ≥1 mg/mg (100 mg/mmol);
4. Estimated glomerular filtration rate (eGFR) calculated using the modified Schwartz formula of ≥60 mL/min/1.73 m².
5. Renal biopsy is optional (if a renal biopsy is performed, cases classified as International Society of Nephropathology (ISKDC) grade ≥IV must be excluded).

Exclusion Criteria:

1. Patients with congenital or acquired immunodeficiency, or those with concurrent tuberculosis, active cytomegalovirus (CMV), Epstein-Barr virus(EBV), hepatitis B, hepatitis C, Human Immunodeficiency Virus(HIV) infection, deep fungal infections, or other active infections;
2. Patients exhibiting the following abnormal laboratory indicators at the time of initial diagnosis: moderate to severe neutropenia (≤1000/μL); moderate to severe anemia (hemoglobin <9.0 g/dL); thrombocytopenia (platelet count <100×10^12/L); or abnormal liver function (Alanine Aminotransferase(ALT), Aspartate Aminotransferase(AST), or bilirubin exceeding 2.5 times the upper limit of normal and persistently elevated for 2 weeks);
3. Patients with a history of tumors or severe cardiovascular, digestive system, hematological, endocrine, or other systemic diseases;
4. Patients with concurrent other urinary system diseases (such as hereditary kidney diseases, etc.);
5. Subjects with severe osteoporosis requiring treatment;
6. Subjects diagnosed with uncontrolled mental illness or intellectual disabilities;
7. Subjects who have received B-cell targeted therapy within the last 6 months;
8. History of major organ transplant or hematopoietic stem cell/cell/bone marrow or kidney transplant;
9. Vaccination with live attenuated vaccines within 1 month prior to treatment;
10. Use of various traditional Chinese medicines for treating kidney diseases during the treatment period (patients who have previously used traditional Chinese medicine can be included, but are strictly prohibited from using it after receiving treatment according to the protocol);
11. Incomplete clinical data.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Collect patients diagnosed with childhood IgA vasculitis nephritis who received treatment with glucocorticoids and/or telitacicept during the treatment period and met the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate of urinary protein [Efficacy] | From enrollment to the 48th week after treatment
  Compared to the baseline, the investigators will assess the proportions of participants with a urine protein-to-creatinine ratio (UPCR) < 0.2 mg/mg (or 20 mg/mmol) or 24-hour urinary protein quantification< 0.2 g/d at weeks 12, 24, and 48 after medication administration.
The rate of change in urinary protein [Efficacy] | From enrollment to the 48th week after treatment
  The investigators will assess the UPCR(mg/mg or mg/mmol) of participants at 12, 24, and 48 weeks after medication administration, comparing the results against the baseline and conducting inter-group comparisons.
The rate of change in urinary protein [Efficacy] | From enrollment to the 48th week after treatment.
  The investigators will assess 24-hour urine protein quantification(g/d) of participants at 12, 24, and 48 weeks after medication administration, comparing the results against the baseline and conducting inter-group comparisons.

SECONDARY OUTCOMES:
Changes in renal function [Safety and Tolerability] | From enrollment to the 48th week after treatment.
  The investigators will assess the changes in estimated glomerular filtration rate (eGFR)(mL/min/1.73m^2) during long-term follow-up, with inter-group comparisons.
Changes in urinary red blood cell count (/μL) [Efficacy] | From enrollment to the 48th week after treatment.
  The investigators will assess the changes in urinary red blood cell count (/μL) during long-term follow-up
Changes in serum immunoglobulin levels [Safety and Tolerability] | From enrollment to the 48th week after treatment.
  The investigators will assess the changes in serum immunoglobulin G、A and M levels (g/L) during long-term follow-up.
Changes in peripheral blood lymphocyte subsets[Efficacy] | From enrollment to the 48th week after treatment.
  The investigators will assess changes in total B and natural killer (TBNK) cells (/μL) during long-term follow-up
Incidence and severity of all adverse events[Safety and Tolerability] | From enrollment to the 48th week after treatment.
  The investigators will assess incidence and severity of all adverse events, including the incidence of infections and hypogammaglobulinemia and the incidence of side effects associated with glucocorticoids.
Cumulative glucocorticoid dosage [Total Dosage] | From enrollment to the 48th week after treatment.
  The investigators will calculate the cumulative glucocorticoid dosage (mg/kg) for each group during the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Mao, Study Chair — Children's Hospital, Zhejiang University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jin Y, Zhu J, Sheng A, Lin Q, Zhao M, He X, Mao J, Fu H. Telitacicept as a BAFF/APRIL dual inhibitor: efficacy and safety in reducing proteinuria for refractory childhood IgA vasculitis nephritis. Pediatr Nephrol. 2025 Aug;40(8):2561-2569. doi: 10.1007/s00467-025-06769-3. Epub 2025 Apr 11. PMID 40214779
- [Result] Wang J, Cui J, Chen J, Liao Y, Yang M, Lin J, Yang X, Zhao B. Telitacicept use in children with IgA vasculitis nephritis: preliminary observations. Pediatr Nephrol. 2025 Sep;40(9):2829-2836. doi: 10.1007/s00467-025-06709-1. Epub 2025 Mar 5. PMID 40042623
- [Result] Liu J, Han X, Jiang X, Gao X, Li G, Fang X, Chen J, Zhai Y, Liu J, Pei Y, Zhang J, Zhu G, Shen Q, Xu H. Efficacy and Safety of Telitacicept as an Add-On Therapy for Refractory Immunoglobulin A Nephropathy or Immunoglobulin A Vasculitis Nephropathy in Children. Kidney Int Rep. 2024 Dec 2;10(3):940-943. doi: 10.1016/j.ekir.2024.11.1363. eCollection 2025 Mar. No abstract available. PMID 40225367
- [Result] Dhillon S. Telitacicept: First Approval. Drugs. 2021 Sep;81(14):1671-1675. doi: 10.1007/s40265-021-01591-1. PMID 34463932
- [Result] Zhang X, Xie X, Shi S, Liu L, Lv J, Zhang H. Plasma galactose-deficient immunoglobulin A1 and loss of kidney function in patients with immunoglobulin A vasculitis nephritis. Nephrol Dial Transplant. 2020 Dec 4;35(12):2117-2123. doi: 10.1093/ndt/gfz151. PMID 31377786
- [Result] Ronkainen J, Nuutinen M, Koskimies O. The adult kidney 24 years after childhood Henoch-Schonlein purpura: a retrospective cohort study. Lancet. 2002 Aug 31;360(9334):666-70. doi: 10.1016/S0140-6736(02)09835-5. PMID 12241872
- [Result] Jauhola O, Ronkainen J, Koskimies O, Ala-Houhala M, Arikoski P, Holtta T, Jahnukainen T, Rajantie J, Ormala T, Turtinen J, Nuutinen M. Renal manifestations of Henoch-Schonlein purpura in a 6-month prospective study of 223 children. Arch Dis Child. 2010 Nov;95(11):877-82. doi: 10.1136/adc.2009.182394. Epub 2010 Sep 18. PMID 20852275
- [Result] Chang WL, Yang YH, Wang LC, Lin YT, Chiang BL. Renal manifestations in Henoch-Schonlein purpura: a 10-year clinical study. Pediatr Nephrol. 2005 Sep;20(9):1269-72. doi: 10.1007/s00467-005-1903-z. Epub 2005 Jun 10. PMID 15947991
- [Result] Watts RA, Hatemi G, Burns JC, Mohammad AJ. Global epidemiology of vasculitis. Nat Rev Rheumatol. 2022 Jan;18(1):22-34. doi: 10.1038/s41584-021-00718-8. Epub 2021 Dec 1. PMID 34853411
- See also: Related Info — https://www.tsgyun.com/official/index.html